CLINICAL TRIAL: NCT05411887
Title: A Non-interventional, Multi Center, Prospective Observational Study to Evaluate the Effect of Improving Systolic Blood Pressure and Low-density Lipoprotein Cholesterol Compared to Conventional Treatments and the Convenience of Taking Medication of Olostar Tab. in Patients With Essential Hypertension and Dyslipidemia.
Brief Title: Study to Evaluate the Effect of Improving Systolic BP and LDL-C Compared to Conventional Treatments and the Convenience of Taking Medication of Olostar Tab
Status: Active, not recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWOS_OLO_004
Record Dates: First submitted 2022-05-19; First posted 2022-06-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hyperlipidemias; Hypertension
MeSH Terms: conditions — Hyperlipidemias; Hypertension | interventions — Rosuvastatin Calcium; Olmesartan Medoxomil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental/ Olostar Tablet: Eligible Subjects who received Olostar Tablet treatment for 24 weeks. Dosage: 10/5mg, 10/10mg, 20/5mg, 20/10mg, 20/20mg, 40/10mg, 40/20mg
  Interventions: Drug: Rosuvastatin, Olmesartan Medoxomil

INTERVENTIONS:
Drug: Rosuvastatin, Olmesartan Medoxomil — Olostar Tablet

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Olostar Tablet on blood pressure and lipid profiles, obtain safety-related information for subgroups that failed to participate in the clinical trials, and to evaluate variables that affect treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. men and women over the age of 19
2. Patients who signed a written consent form to participate in the study
3. Patients who are eligible for Olostar tablet prescription according to domestic permission

Exclusion Criteria:

1. A person who falls under "2. Do not administer to the following patients" among the precautions for use in the user manual
2. Patients in hospital (hospitals only; nursing care facilities can be recruited)
3. A person who has been administered the study target drug or is being administered at the time of recruitment within 6 months based on the date of the study contract

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3000 subjects is a sufficient number to produce a meaningful model considering discriminant analysis and regression analysis that will be conducted in the secondary evaluation
Sampling Method: Probability Sample
Enrollment: 2845 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
absolute change and rate of change in low-density lipoprotein cholesterol (LDL-C) | 24 weeks
  Evaluation of absolute change and rate of change in low-density lipoprotein cholesterol (LDL-C) compared to baseline
absolute change and rate of change in systolic and diastolic blood pressure | 24 weeks
  Evaluation of absolute change and rate of change in systolic and diastolic blood pressure compared to baseline

SECONDARY OUTCOMES:
Proportion of subjects who achieved both general hypertension treatment goals and blood low-density lipoprotein cholesterol (LDL-C) treatment goals | 24 weeks
  Proportion of subjects who achieved both general hypertension treatment goals and blood low-density lipoprotein cholesterol (LDL-C) treatment goals assessed 6 months after administration of Olosta tablets
LDL-C treatment goal achievement rate | 24 weeks
  LDL-C treatment goal achievement rate at 24 weeks
Blood pressure treatment goal achievement rate | 24 weeks
  Blood pressure treatment goal achievement rate at 24 weeks
Proportion of subjects who decreased systolic blood pressure by 20 mmHg and diastolic blood pressure by 10 mmHg | 24 weeks
  Proportion of subjects who decreased systolic blood pressure by 20 mmHg and diastolic blood pressure by 10 mmHg at 24 weeks
Olostar tablet compliance | 24 weeks
  Olostar tablet compliance at 24 weeks
Olostar tablet dose change | 24 weeks
  Olostar tablet dose change: ① Proportion of subjects by initial dose, ② Average number of dose changes, ③ Proportion of subjects by dose at the end at 24 weeks
Olostar Tablet persistence | 24 weeks
  Olostar Tablet persistence: ① persistence rate; ② Median time to discontinuation; ③ Evaluation of reasons for suspension
Evaluation of compliance | 24 weeks
  Evaluation of compliance with therapeutic lifestyle improvement (eating habits and amount of exercise)
Assessment of Variables Influencing the Simultaneous Achievement of General | 24 weeks
  Assessment of Variables Influencing the Simultaneous Achievement of General Treatment Goals for Hypertension and Low-Density Lipoprotein Cholesterol (LDL-C) Treatment Goals and the Creation of a Predictive Model at 24 weeks
Evaluation of variables affecting the frequency and severity of safety (adverse drug reactions, etc.) | 24 weeks
  Evaluation of variables affecting the frequency and severity of safety (adverse drug reactions, etc.) at 24 weeks
Evaluation of variables affecting compliance and persistence with Olostar tablets | 24 weeks
  Evaluation of variables affecting compliance and persistence with Olostar tablets at 24 weeks
Evaluation of convenience of taking Olostar tablets | 24 weeks
  Evaluation of convenience of taking Olostar tablets at 24 weeks
Actual incidence of adverse events, adverse drug reactions, and serious adverse events in subjects receiving Olostar tablets | 24 weeks
  Actual incidence of adverse events, adverse drug reactions, and serious adverse events in subjects receiving Olostar tablets at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JaeWon Oh, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No